CLINICAL TRIAL: NCT04701125
Title: Selective Head-neck Cooling Following Concussion Shortens Return-to-play in Ice Hockey Players
Brief Title: Medical Cooling of Ice Hockey Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BC123122334
Record Dates: First submitted 2020-12-28; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Sports-related Concussions, Selective Head-neck Cooling, Return to Play

STUDY DESIGN:
Intervention Model Description: Twenty-eight teams from the elite ice hockey leagues for males in Sweden were invited to participate in the study. Participating teams were given the option to be in the study group (receiving selective head-neck cooling after SRC) or the control group (standard SRC management). Any player with a suspected or diagnosed concussion was immediately removed from practice or game participation for further evaluation. Concussion diagnosis was established using the concussion in the sports consensus statement. At the time of SRC, any presence of "red flags" mandated the player to be taken to the hospital. As soon as the diagnosis of SRC was established the player was included in the study and players in the intervention teams were treated by selective head-neck cooling system for a minimum of 30 minutes. The primary endpoint of the study was the time (in days) from concussion until returning to full practice or game.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Players receive selective head-neck cooling after concussion
  Interventions: Device: selective head-neck cooling using PolarCap system
- control group (No Intervention): Players receive the standard sport-related concussion management

INTERVENTIONS:
Device: selective head-neck cooling using PolarCap system — Players receiving selective head-neck cooling after SRC
  Arms: Study group

SUMMARY:
The incidence of Sports-related concussions (SRCs) has risen in recent years, not least in ice hockey, and available treatment options are limited. Here, we addressed the hypotheses that immediate controlled head- and neck cooling could hasten return-to-play in a Swedish cohort of concussed professional ice hockey players. Over three seasons, 15 teams used either immediate head- and neck cooling or standard management for SRC. All players (81) followed the same return-to-play management protocol.

DETAILED DESCRIPTION:
Sports-related concussions (SRCs) are a growing health concern, since they may lead to persistent symptoms and, particularly if repeated, to e.g. depression, accelerated dementia onset, and development of chronic traumatic encephalopathy. Here, we addressed the hypotheses that immediate controlled head- and neck cooling could hasten return-to-play in a Swedish cohort of concussed professional ice hockey players. Over three seasons, 15 teams used either immediate head- and neck cooling or standard management for SRC. All players followed the same return-to-play management protocol. Using a baseline questionnaire, no difference in the number of previous SRCs between groups was observed. In total, 92 SRCs were recorded. Eleven players did not complete the study protocol, and thus 81 players were included. Of these, 29 were treated by immediate selective head- and neck cooling for ≥ 30 min, and 52 controls received standard acute SRC management.

ELIGIBILITY:
Inclusion Criteria:

* Elite ice hockey players diagnosed by a team physician to have suffered a sports-related concussion. Selective head-neck cooling following the concussion. Duration of cooling a minimum of 45 minutes.

Exclusion Criteria:

* Presence of red flags (loss of consciousness, seizure, worsening headache, repeated vomiting, focal neurological deficits, neck pain, tingling in arms). Inability to tolerate cooling for a minimum of 30 minutes. Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
return-to-play | two weeks
  The primary endpoint of the study was time (in days) from concussion until returning to full practice or game

CONTACTS AND LOCATIONS:
Locations (1):
- University, Lund, Sweden